CLINICAL TRIAL: NCT00528489
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of PENNVAX-B (Gag, Pol, Env) Given Alone, With IL-12 DNA, or With a Dose Escalation of IL-15 DNA, in Healthy, HIV-1-uninfected Adults Participants
Brief Title: Safety and Effectiveness of PENNVAX-B Vaccine Alone, With Il-12, or IL-15 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 070; 10490 (Registry Identifier: DAIDS ES Registry ID)
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; DNA Plasmid Vaccine; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-12; Interleukin-15

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Experimental): PENNVAX-B with 0.8 mg IL-15 administered in both deltoids at Months 0, 1, 3, and 6
  Interventions: Biological: PennVax B; Biological: IL-15
- 2 (Experimental): PENNVAX-B administered alone in both deltoids at Months 0, 1, 3, and 6
  Interventions: Biological: PennVax B
- 3 (Experimental): PENNVAX-B administered alone in both deltoids at Months 0, 1, 3, and 6
  Interventions: Biological: PennVax B; Biological: IL-12
- 4 (Experimental): PENNVAX-B with 2 mg IL-15 injected into both deltoids at Months 0, 1, 3, and 6
  Interventions: Biological: PennVax B; Biological: IL-15

INTERVENTIONS:
Biological: PennVax B — DNA vaccine containing the HIV genes Gag, Pol, and Env
Biological: IL-12 — Cytokine injection
  Arms: 3
Biological: IL-15 — Cytokine injection
  Arms: 1; 4

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and immune response to the DNA HIV vaccine, PENNVAX-B alone, in combination with IL-12, or with 2 different doses of IL-15.

DETAILED DESCRIPTION:
A vaccine that is effective against multiple strains of HIV remains the best option for preventing the spread of HIV. Plasmid DNA vaccines are inexpensive and easy to construct. When DNA vaccines are administered in combination with cytokines, such as IL-12 or IL-15, the immune response to the vaccine is increased. The purpose of this study is to determine the safety and tolerability of the DNA plasmid vaccine, PENNVAX-B when administered alone, or with IL-12 or IL-15 DNA adjuvants. The most effective and safe dose of IL-15 will also be determined during this study.

This study will last approximately 12 months. Participants will be randomly assigned to one of four groups. Group 1 will receive an injection of PENNVAX-B combined with 0.8 mg IL-15 in each deltoid or placebo. Group 2 will receive an injection of PENNVAX-B alone or placebo. Group 3 will receive an injection of PENNVAX-B combined with IL-12 in each deltoid or placebo. Group 4 will receive PENNVAX-B combined with 2 mg IL-15 or placebo. Injections will occur at study entry, Months 1, 3, and 6. Additional study visits will occur on Days 14, 42, 98, 182, 273, and 364. At these visits a brief physical, blood collection, interview, and risk reduction counseling will occur. At some visits HIV testing, urine collection, and pregnancy tests will also occur.

As of 05/30/08, participants will be enrolled into Groups 3 and 4 at a limited pace to allow for additional safety reviews for the first few participants in these groups. Additionally, safety data will be reviewed for Groups 1 and 2 to determine whether the remainder of participants in Groups 2, 3, and 4 will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 and -2 uninfected
* Willing to receive HIV test results
* Good general health
* Certain laboratory values within normal range or with site physician approval
* Negative for Hepatitis B surface antigen
* Negative Hepatitis C test
* Willing to use acceptable methods of contraception

Exclusion Criteria:

* HIV vaccines or placebos in prior HIV trial. Participants who can provide documentation that they received a placebo in a prior HIV trial may be eligible.
* Immunosuppressive medications within 168 days prior to first study vaccination. Participants using corticosteroid nasal spray for allergies or topical corticosteroids for mild, uncomplicated dermatitis are not excluded.
* Blood products within 120 days prior to first study vaccination
* Receipt of immunoglobulin within 60 days prior to first vaccination
* Live attenuated vaccines within 30 days prior to first study vaccination
* Any vaccine that is not a live attenuated vaccine within 14 days prior to first study vaccination
* Investigational research agents within 60 days prior to first study vaccination
* Current anti-tuberculosis (TB) preventive therapy or treatment clinically significant medical condition, abnormal physical exam findings, abnormal laboratory results, or past medical history that may affect current health. More information about this criterion can be found in the protocol.
* Any medical, psychiatric, social, occupational, or other condition or responsibility that in the opinion of the investigator would interfere with the study. More information about this criterion can be found in the protocol.
* Allergy to amide-type local anesthetics
* Serious adverse reactions to vaccines
* Autoimmune disease or immunodeficiency
* Active syphilis infection. Participants who have been fully treated for syphilis over 6 months prior to study entry are not excluded.
* Asthma other than mild, well-controlled asthma. More information on this criterion can be found in the protocol.
* Type 1 or type 2 diabetes mellitus. Participants with histories of isolated gestational diabetes are not excluded.
* Thyroidectomy or thyroid disease requiring medication during the 12 months prior to study entry
* Accumulation of fluid in the blood vessels (angioedema) within 3 years prior to study entry if episodes are considered serious or have required medication in the 2 years prior to study entry
* Uncontrolled hypertension
* Body Mass Index of 40 or greater OR of 35 or greater if certain other criteria apply. More information about these criteria can be found in the protocol
* Bleeding disorder
* Cancer. Participants with surgically removed cancer that is unlikely to recur are not excluded.
* Seizure disorder
* Absence of the spleen
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety data including local and systemic reactogenicity sign and symptoms, laboratory measures of safety, and adverse and serious adverse events | Throughout study
Safety data from Groups 1 and 4 | Throughout study

SECONDARY OUTCOMES:
HIV-1 specific interferon gamma ELISpot and/or intracellular cytokine staining T cell response | 2 weeks after 3rd and 4th vaccinations
HIV-1 specific neutralizing and binding antibody assays | 2 weeks after 3rd and 4th vaccinations

CONTACTS AND LOCATIONS:
Overall Officials: Scott Parker, MD, Study Chair — HVTN, FHCRC
Locations (8):
- United States (8):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - Brigham and Women's Hosp. CRS, Boston, Massachusetts
  - NY Blood Ctr./Union Square CRS, New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - NY Blood Ctr./Bronx CRS, The Bronx, New York
  - 3535 Market Street CRS, Philadelphia, Pennsylvania
  - Vanderbilt Vaccine CRS, Nashville, Tennessee

REFERENCES:
- [Background] Johnston MI, Fauci AS. An HIV vaccine--evolving concepts. N Engl J Med. 2007 May 17;356(20):2073-81. doi: 10.1056/NEJMra066267. No abstract available. PMID 17507706
- [Background] Ogawa H, Ueno M, Uchibori H, Matsumoto I, Seno N. Direct carbohydrate analysis of glycoproteins electroblotted onto polyvinylidene difluoride membrane from sodium dodecyl sulfate-polyacrylamide gel. Anal Biochem. 1990 Nov 1;190(2):165-9. doi: 10.1016/0003-2697(90)90175-9. PMID 1705391
- [Background] McBurney SP, Ross TM. Developing broadly reactive HIV-1/AIDS vaccines: a review of polyvalent and centralized HIV-1 vaccines. Curr Pharm Des. 2007;13(19):1957-64. doi: 10.2174/138161207781039841. PMID 17627529
- [Derived] Jin X, Morgan C, Yu X, DeRosa S, Tomaras GD, Montefiori DC, Kublin J, Corey L, Keefer MC; NIAID HIV Vaccine Trials Network. Multiple factors affect immunogenicity of DNA plasmid HIV vaccines in human clinical trials. Vaccine. 2015 May 11;33(20):2347-53. doi: 10.1016/j.vaccine.2015.03.036. Epub 2015 Mar 25. PMID 25820067
- See also: Click here to learn more about the HIV Vaccine Trials Network — http://www.hvtn.org